CLINICAL TRIAL: NCT04209933
Title: Comparison of Efficacy of Bismuth Potassium Citrate, Pectin Bismuth Capsules, and Pectin Bismuth Granules in the Treatment of Helicobacter Pylori (Hp) First-line Quadruple Regimen: a Multicenter, Randomized, Prospective, Comparative Clinical Trial
Brief Title: Helicobacter Pylori Eradication With Different Bismuth Quadruple Therapies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20192146-C-1
Record Dates: First submitted 2019-12-13; First posted 2019-12-24 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Gastric Cancer; Helicobacter Pylori Infection; Bismuth
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bismuth potassium citrate containing quadruple therapy (Active Comparator): Bismuth potassium citrate 220 mg,rabeprazole 10 mg, amoxicillin 1000mg, and clarithromycin 500 mg by mouth,twice daily for 14 days.
  Interventions: Drug: Bismuth potassium citrate containing quadruple therapy; Drug: Colloidal pectin bismuth capsules containing quadruple therapy; Drug: Colloidal pectin bismuth particles A quadruple therapy; Drug: Colloidal pectin bismuth particles B quadruple therapy
- Colloidal pectin bismuth capsules containing quadruple therapy (Active Comparator): Colloidal pectin bismuth capsules 200 mg,rabeprazole 10 mg, amoxicillin 1000mg, and clarithromycin 500 mg by mouth,twice daily for 14 days.
  Interventions: Drug: Bismuth potassium citrate containing quadruple therapy; Drug: Colloidal pectin bismuth capsules containing quadruple therapy; Drug: Colloidal pectin bismuth particles A quadruple therapy; Drug: Colloidal pectin bismuth particles B quadruple therapy
- Colloidal pectin bismuth particles A quadruple therapy (Active Comparator): Colloidal pectin bismuth particles 150 mg,rabeprazole 10 mg, amoxicillin 1000mg, and clarithromycin 500 mg by mouth,twice daily for 14 days.
  Interventions: Drug: Bismuth potassium citrate containing quadruple therapy; Drug: Colloidal pectin bismuth capsules containing quadruple therapy; Drug: Colloidal pectin bismuth particles A quadruple therapy; Drug: Colloidal pectin bismuth particles B quadruple therapy
- Colloidal pectin bismuth particles B quadruple therapy (Active Comparator): Colloidal pectin bismuth particles 300 mg,rabeprazole 10 mg, amoxicillin 1000mg, and clarithromycin 500 mg by mouth,twice daily for 14 days.
  Interventions: Drug: Bismuth potassium citrate containing quadruple therapy; Drug: Colloidal pectin bismuth capsules containing quadruple therapy; Drug: Colloidal pectin bismuth particles A quadruple therapy; Drug: Colloidal pectin bismuth particles B quadruple therapy

INTERVENTIONS:
Drug: Bismuth potassium citrate containing quadruple therapy — Bismuth potassium citrate:given for 14 days at a dose of bismuth potassium citrate 220 mg 0 BID,rabeprazole 10 mg BID, amoxicillin 1000 mg BID, and clarithromycin 500 mg BID
Drug: Colloidal pectin bismuth capsules containing quadruple therapy — Bismuth potassium citrate:given for 14 days at a dose of Colloidal pectin bismuth capsules 200 mg 0 BID,rabeprazole 10 mg BID, amoxicillin 1000 mg BID, and clarithromycin 500 mg BID
Drug: Colloidal pectin bismuth particles A quadruple therapy — Bismuth potassium citrate:given for 14 days at a dose of Colloidal pectin bismuth particles 150 mg BID,rabeprazole 10 mg BID, amoxicillin 1000 mg BID, and clarithromycin 500 mg BID
Drug: Colloidal pectin bismuth particles B quadruple therapy — Bismuth potassium citrate:given for 14 days at a dose of Colloidal pectin bismuth particles 300 mg BID,rabeprazole 10 mg BID, amoxicillin 1000 mg BID, and clarithromycin 500 mg BID

SUMMARY:
This study aims to compare efficacy and safety of bismuth-containing quadruple therapy（with rabeprazole amoxicillin clarithromycin）of different kinds of bismuth（Bismuth potassium citrate, pectin bismuth capsules, pectin bismuth particles）in H. pylori first-line eradication. It is hypothesized that different bismuth containing quadruple therapies have comparable eradication efficacy and safety. Patients with confirmed H. pylori positive status will be randomized to one of the treatments described above. At week 2and 6 follow-up visits, a urea breath test(UBT) will be performed to confirm eradication.

DETAILED DESCRIPTION:
The study will include three phases: screening, treatment and follow-up.Screening: this phase will last a maximum of 28 days and subjects eligibility will be evaluated after informed consent signature. Endoscopy and Urea Breath test will be performed in addition to the baseline routine evaluations.Treatment: Subjects are randomly assigned to treatment and will be treated for 14 days. A randomization visit will take place on Day 0 and an end-of-treatment visit will take place between day 12 and 14.Follow-up: includes two visits. approximately 14 days of treatment and 28 days after the end of treatment. Eradication of H. Pylori will be confirmed through urea breath test(UBT).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18~75,both gender.
* Patients with upper gastrointestinal symptoms and with documented H.pylori infection.
* Patients are willing to receive eradication treatment.
* Women are eligible if they are not pregnant or nursing, and if they are of childbearing potential they are required to use medically acceptable contraception for the duration of the study and 30 days thereafter.

Exclusion Criteria:

* Patients are excluded if they have previously used antibiotics to eradicate adequately recorded infection with H. pylori.
* Contraindications to study drugs.
* Substantial organ impairment, severe or unstable cardiopulmonary or endocrine disease.
* Constant use of anti-ulcer drugs ( including taking proton-pump.inhibitors(PPI) within 2 weeks before the [13C] urea breath test),antibiotics or bismuth complexes (more than 3 times /1 month before screening).
* Patients were diagnosed with gastroduodenal ulcer and MALTlymphoma.
* Pregnant or lactating women.
* Underwent upper gastrointestinal Surgery.
* Patients with Barrett esophageal or highly atypical hyperplasia, have symptom of dysphagia.
* Evidence of bleeding or iron efficiency anemia.- Page 3 of 4 [DRAFT] -
* A history of malignancy.
* Drug or alcohol abuse history in the past 1 year.
* Systemic use of corticosteroids, non steroidal anti-inflammatory drugs,anticoagulants, platelet aggregation inhibitors (except the use of aspirin for less than 100 mg/d).
* Patients who has psychological problem or poor compliance.
* Enrolled in other clinical trials in the past 3 months.
* Refuse to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
helicobacter pylori eradication | 28 days after treatment]
  The primary end point of this study is H.pylori eradication,established by negative [13C] urea breath test 28 days after the end of eradication.

SECONDARY OUTCOMES:
symptoms effective rates | 14 days of treatment, and 28 days after treatment
  symptoms effective rates Evaluation effective rate of symptoms 2 weeks of treatment and 4 weeks after the end of treatment. Symptom effective rate =#total score before treatment - total score after treatment#/total score before treatment x100%. Total score = frequency + severity.Frequency score is calculated by all the frequency of heartburn, reflux, abdominal pain, and flatulence. Severity is accumulated by the degree of symptoms described above, which is divided to 4 degree as 0 presenting none, and 3presenting most severe

OTHER OUTCOMES:
adverse events | 14 days of treatment, and 28 days after treatment
  Participants with Adverse Events as a Measure of Safety and Tolerability.The common side effects of the study include headache, dizziness, skin rash, other gastrointestinal disorders, pyrexia, cough and back pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao Y, Zhang J, Liu Y, Zhang L, Wang L, Wang J, Qi Y, Lv H, Liu J, Huo L, Wei X, Shi Y. The efficacy and safety of different bismuth agents in Helicobacter pylori first-line eradication: A multicenter, randomized, controlled clinical trial. Medicine (Baltimore). 2021 Dec 17;100(50):e27923. doi: 10.1097/MD.0000000000027923. PMID 34918639